CLINICAL TRIAL: NCT01427062
Title: Effects of an Innovative Balance Training Programme in Enhancing Postural Control and Reducing Falls in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Margaret Kit Yi Mak, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PD-001
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Parkinson's Disease
Keywords: parkinson's disease; balance; anticipatory postural adjustment; componsatory postural adjustment; falls
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- anticipatory and compensatory postural control training (Experimental): Subjects in the experimental group were trained the speed and amplitude of anticipatory postural adjustment during fall-prone activities and postural response to perturbation during walking. Training was provided with preparatory cues, computerized machines and treadmill.
  Interventions: Other: experimental
- strength-focused training (Active Comparator): Subjects in control group were provided with strength training of leg muscles using machines and during functional activities.
  Interventions: Other: control

INTERVENTIONS:
Other: experimental — Subjects in the experimental group were trained the speed and amplitude of anticipatory postural adjustment during fall-prone activities and postural response to perturbation during walking. Training was provided with preparatory cues, computerized machines and treadmill.
  Arms: anticipatory and compensatory postural control training
Other: control — Subjects in control group were provided with strength training of leg muscles using machines and during functional activities.
  Arms: strength-focused training

SUMMARY:
Falling is a complex and most disabling feature for patients with Parkinson's disease (PD). Previous studies suggested that falls in patients with PD are related to postural instability characterized by deficits in anticipatory postural adjustment (APA) for postural orientation in walking and standing and inadequate postural response to perturbation. The present study developed an innovative balance treatment with focus of anticipatory and compensatory postural control and examined its effects on enhancing balance and gait performance and decreasing fall rate in people with PD.

DETAILED DESCRIPTION:
Participants: Forty-two eligible subjects with PD were randomly allocated into balance with focus of anticipatory and compensatory postural control (EXP) or control (CON) group with strength-focused training, with 26 subjects in each group.

Methods: Subjects in the EXP group were trained the speed and amplitude of anticipatory postural adjustment during stepping and walking and postural response to perturbation during walking. Subjects In the CON group were trained to improve the strength of lower limb muscles. Treatment period in both groups lasted for 12 weeks, which consisted of 4-week laboratory-based training (phase 1), 4-week home-based exercise (phase 2) and final 4-week laboratory-based training (phase 3). Outcome measures included reaction time(RT), movement velocity (MV) and endpoint excursion (EPE) of limit-of-stability test, one-leg-stance (OLS) time, gait velocity, stride length (SL), cadence, and fall rate. All tests were conducted for 6 time intervals including baseline, after each training phase, at 3-month follow-up and at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as parkinson's disease
2. 45 years old or above
3. stable on anti-parkinsonian medications for at least 6 weeks prior to entry into the study, which will remain unchanged for the duration of the study
4. able to walk a 10 meter distance at least 3 times with or without walking aids independently
5. at stage 2 or 3 of the Hoehn and Yahr staging
6. able to provide informed consent

Exclusion Criteria:

1. neurological conditions other than PD
2. uncompensated cardiovascular disease
3. less than 23 score on the Mini-Mental State examination,
4. History of fracture or recent musculoskeletal disorders in back or lower limbs which would interfere with the balance during exercise and daily activities
5. visual disturbance or vestibular dysfunction limiting locomotion or balance
6. participation in other balance-related training program more than one time per week

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
reaction time of limits of stability test | One year
one-leg-stance time | one year
pull test | one year
  it reflects the ability of compensatory postural control in patients with Parkinson's disease
fall rate | previous one year before baseline assessment, each following one month for 3-month of training and 12-month of follow-up
movement velocity of limit of stability test | one year
end point excursion of limits of stability test | One year

SECONDARY OUTCOMES:
Unified Parkinson's Disease rating scale- motor examination subscale | one year
  it reflects motor impairment of patients with Parkinson's disease
Gait velocity | one year
Stride length | One year
Cadence | One year

CONTACTS AND LOCATIONS:
Overall Officials: Xia SHEN, PHD candidate, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Locations (1):
- the Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886